CLINICAL TRIAL: NCT06466655
Title: Accelerated Vascular Aging in Midlife as a Mechanism Linking Daily Stress to Cognitive Decline
Brief Title: Daily Stress and Vascular Function in Midlife as a Risk Factor for Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2056784; 2P20GM113125 (NIH)
Record Dates: First submitted 2024-06-04; First posted 2024-06-20 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-05

CONDITIONS: Middle-aged Adults; Major Depressive Disorder
Keywords: intradermal microdialysis; microvascular function; endothelium-dependent dilation; nitric oxide; stress; cognitive function
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- middle-aged healthy adults (Active Comparator): middle-aged healthy adults
  Interventions: Drug: MitoTempol; Drug: Lactated Ringer's (control)
- middle-aged adults with major depressive disorder (Experimental): middle-aged adults with major depressive disorder
  Interventions: Drug: MitoTempol; Drug: Lactated Ringer's (control)

INTERVENTIONS:
Drug: MitoTempol — One intradermal microdialysis probes will be perfused with MitoTempol (0.5 mM) during a standard local skin heating protocol.
Drug: Lactated Ringer's (control) — One intradermal microdialysis probes will be perfused with lactated Ringer's (control) during a standard local skin heating protocol.

SUMMARY:
The goal of this pilot clinical trial is to begin to understand how day-to-day stress affects cardiovascular health and brain function in middle-aged adults. The main question aims to answer is whether the link between daily stress and vascular dysfunction is a potential mechanism of increased risk for future cognitive decline. Participants will complete a 15-day testing cycle. During this cycle, participants will complete daily assessments of stress using an online survey tool for 14-consecutive days. On the last day of each cycle, vascular function will be assessed during a laboratory visit.

DETAILED DESCRIPTION:
Because of global demographic trends toward increasingly older populations, there is an urgent need to identify the mechanistic underpinnings of modifiable risk factors for age-related chronic disease risk starting in midlife in order to establish novel biological targets for therapeutic intervention strategies that can be implemented earlier in the aging trajectory and prior to clinically detectable declines in function. Major depressive disorder (MDD) is the leading cause of disability and disease burden in midlife. Accordingly, the long-term goal is to determine whether and to what extent mitochondrial reactive oxygen species (mtROS)-induced impairments in peripheral endothelium-dependent dilation (EDD) explain how daily stress impacts 'real-world' cognitive function in middle-aged adults with MDD. As a necessary first step, the objective of this pilot trial is to examine the degree to which mtROS contributes to nitric oxide-dependent EDD in middle-aged adults with major depressive disorder.

A small community sample of cognitively unimpaired middle-aged males and females with and without MDD (n=20; 40-55 yrs) will be recruited. Participants will be recruited from New Castle County, Delaware (DE) and surrounding regions and will be representative of the sex/ethnic/racial population of DE. After providing verbal and written consent, all participants will undergo a clinical exam for signs and symptoms of chronic disease by clinical nursing staff. This will include a complete health history (females will also complete a gynecological history, including a 3-mo menstrual cycle recall), physical exam (anthropometry, resting hemodynamics, and a 12-lead electrocardiogram), and basic blood biochemistry (complete blood count, lipid profile, renal function, electrolytes, HbA1c, fasting glucose and insulin).

Ambulatory Assessment Protocol (Days 1-14): Daily stress processes will be assessed each day during the last daily assessment using an adapted version of the Daily Inventory of Stressful Events (DISE; ~8 min). Daily cognitive function will be assessed in multiple domains (subjective and objective).

Laboratory Assessment of Peripheral Endothelial Function (Day 15): Microvascular endothelial function will be assessed using intradermal microdialysis coupled with laser Doppler flowmetry. Two intradermal microdialysis probes (CMA Linear 31 probe, 55 kDa) will be inserted into the dermal layer of the ventral forearm and perfused with either lactated Ringer's solution (control) or MitoTempol (0.5 mM) to scavenge mitochondrial-derived superoxide. Red cell flux will be continuously measured via integrated laser Doppler flowmeters. Mean arterial pressure will be measured via brachial auscultation every 4 min. A standard local heating protocol will be used to elicit EDD and the NO-dependent portion of this response will be determined pharmacologically, as previously described.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 40-55 yrs
* Absence of objective cognitive impairment (≥26 on the Montreal Cognitive Assessment)
* Absence of diagnosed or unstable neurocognitive, cardiovascular, metabolic, renal, hepatic, autonomic, autoimmune, or dermatological diseases, as determined by medical history, physical examination, blood chemistries, and 12-lead resting electrocardiogram
* Participants must have a level of understanding of the English language sufficient to provide informed consent and to agree to all tests and procedures, as well as the capacity and willingness to attend all study related visits and to comply with the study protocol

Exclusion Criteria:

Subjects will be excluded at the discretion of the PI/collaborating clinicians or for any of the following reasons:

* <40 or >55 yrs
* Psychiatric illness aside from MDD (e.g., bipolar disorder, schizophrenia, eating disorders), assessed by the MINI and self-report
* Objective cognitive impairment (<26 on the Montreal Cognitive Assessment)
* Diagnosed or unstable neurocognitive, cardiovascular, metabolic, renal, hepatic, autonomic, autoimmune, or dermatological diseases
* Current or recent use (within 8 wks) of medications that alter cardiovascular function or psychoactive/psychopharmacological drugs
* Body mass index ≥35 kg/m2
* Resting systolic BP ≥140 mmHg
* HbA1c ≥5.7%
* Direct low-density lipoprotein ≥160mg/dl
* Tobacco use (including electronic cigarettes)
* Females who are pregnant, breastfeeding, or planning to become pregnant; female subjects of child-bearing age must have a negative urine pregnancy test on the day of all experimental visits
* Current or past use of hormone replacement therapy
* Allergy to study drugs or pharmacological agents

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jody Greaney, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
Analysis scripts will be shared via the Open Science Framework.
Supporting Information: Analytic Code
Time Frame: Analysis scripts will shared at the time of the associated publication.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We have IRB approval for additional assessments which are being used to address to separate hypotheses and are not contained under this clinical trial.
Groups:
- Middle-aged Healthy Adults (HA): cognitively intact healthy middle-aged adults
- Middle-aged Adults With Major Depressive Disorder (MDD): cognitively intact middle-aged adults with major depressive disorder
Period: Overall Study
Arm/Group | Middle-aged Healthy Adults (HA) | Middle-aged Adults With Major Depressive Disorder (MDD)
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Middle-aged Healthy Adults: cognitively intact healthy middle-aged adults
- Middle-aged Adults With Major Depressive Disorder: cognitively intact middle-aged adults with major depressive disorder
- Total: Total of all reporting groups
Arm/Group | Middle-aged Healthy Adults | Middle-aged Adults With Major Depressive Disorder | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (4) | 51 (4) | 51 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 6 | 6 | 12
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
body mass index [Mean (Standard Deviation); unit: kilograms per meter-squared] | 23.8 (2.3) | 26.0 (3.8) | 24.9 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Nitric Oxide (NO)-Mediated Endothelium-dependent Dilation (EDD)
Description: NO-mediated EDD will be calculated as the relative difference (%) in dilation from the local heating-induced plateau to the post-L-NAME plateau after scavenging mitochondrial-derived superoxide
Time Frame: Day 15 following a standard local heating protocol, an average of 4 hours during the 15-day cycle
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Middle-aged Healthy Adults: cognitively intact middle-aged healthy adults
Arm/Group | Middle-aged Healthy Adults | Middle-aged Adults With Major Depressive Disorder
Number analyzed (Participants) | 9 | 8
percentage | 70 (9) | 74 (15)
Statistical Analysis 1: Comparison: Middle-aged Healthy Adults vs Middle-aged Adults With Major Depressive Disorder; Test type: Equivalence; p > 0.05, t-test, 2 sided

2. Secondary Outcome: Local Heating-induced Endothelium-dependent Dilation (EDD)
Description: Local heating-induced EDD will be calculated as the relative difference (%) in dilation during the local heating-induced plateau compared to baseline after scavenging mitochondrial-derived superoxide
Time Frame: Day 15 following a standard local heating protocol, an average of 4 hours during the 15-day cycle
Population: middle-aged adults
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Middle-aged Healthy Adults | Middle-aged Adults With Major Depressive Disorder
Number analyzed (Participants) | 9 | 8
percent | 89 (10) | 93 (11)
Statistical Analysis 1: Comparison: Middle-aged Healthy Adults vs Middle-aged Adults With Major Depressive Disorder; Test type: Equivalence; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: only during 15 days of the testing cycle
Groups:
- Middle-adults With Major Depressive Disorder: cognitively intact middle-aged adults with major depressive disorder
Arm/Group | Middle-aged Healthy Adults | Middle-adults With Major Depressive Disorder
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT06466655/Prot_SAP_ICF_000.pdf